CLINICAL TRIAL: NCT06113809
Title: Phase Ib Trial Evaluating the Combination of CDK4 Inhibitor With Immunotherapy in Patients With Sarcoma
Brief Title: Palbociclib and Pembrolizumab in Sarcoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: John Rieth (Other)
Responsible Party: Sponsor-Investigator, John Rieth, Clinical Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202305133
Record Dates: First submitted 2023-10-16; First posted 2023-11-02 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — palbociclib; pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is a single-arm open-label window of opportunity clinical study assessing the impact of pre-treatment with palbociclib
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination of Palbociclib with Pembrolizumab (Experimental): Palbociclib given for 2 weeks following a pre-treatment ultrasound guided biopsy used to establish an immunological baseline of the tumor microenvironment. After the conclusion of palbociclib therapy, a post-treatment biopsy will be performed to assess the impact of palbociclib on the tumor microenvironment; pembrolizumab will be started the same day as the second biopsy. After 2 doses of pembrolizumab, a third (optional) biopsy could be performed.
  Interventions: Drug: Palbociclib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Palbociclib — Palbociclib is a CDK4/6 inhibitor.
  Palbociclib, 125 mg, (pediatric dose 75mg/m2 up to 125mg) daily for 21 days out of every 28 days, PO (orally) starting 14 days prior to Pembrolizumab
Drug: Pembrolizumab — Pembrolizumab is a PD-1 blocking antibody.
  Given 14 days following Palbociclib: Pembrolizumab, 200 mg, once every three weeks, intravenously (IV)

SUMMARY:
This is a single-arm open-label window of opportunity clinical study assessing the impact of pre-treatment with palbociclib in patients with soft tissue sarcomas for which PD-1 inhibitors are approved (includes undifferentiated pleomorphic sarcoma, myxofibrosarcoma, angiosarcoma, pleomorphic rhabdomyosarcoma, pleomorphic liposarcoma, or alveolar soft part sarcoma).

DETAILED DESCRIPTION:
Patients will be given palbociclib for 2 weeks following a pre-treatment ultrasound guided biopsy used to establish immunological baseline of the tumor microenvironment. After 2 weeks of palbociclib therapy, a second biopsy will be performed to assess the impact of palbociclib on the tumor microenvironment. Pembrolizumab will be started the same day as the second biopsy. After 2 doses of pembrolizumab, a third (optional) biopsy may be performed if the subject consents. At 8 weeks of therapy disease response will be assessed as per standard of care.

ELIGIBILITY:
Inclusion Criteria

A potential subject must meet all the following inclusion criteria to be eligible to participate in the study:

* Male or female patients aged > or = 12 years old
* ECOG Performance Status of < or = 2
* Any patient with the diagnosis of locally advanced, unresectable or metastatic sarcoma for which PD-1 inhibitors are approved (undifferentiated pleomorphic sarcoma, myxofibrosarcoma, angiosarcoma, pleomorphic rhabdomyosarcoma, pleomorphic liposarcoma, alveolar soft part sarcoma) who have progressed on at least 1 prior line of therapy. Prior immunotherapy treatment is allowed, including prior treatment with a PD-1 inhibitor.
* Patients with no known CNS disease, except for treated brain metastasis. Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing treatment for dexamethasone (as ascertained by clinical examination and brain imaging) during the screening period. Stable dose of anticonvulsants is allowed. Treatment for brain metastases may include whole brain radiotherapy, radiosurgery, or a combination as deemed appropriate by the treating physician. Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day 1 will be excluded.
* Ability to understand and the willingness to sign a written informed consent or assent in case of patients < 18 years old.

Exclusion Criteria

A potential subject who meets any of the following exclusion criteria is ineligible to participate in the study:

* Lab values in the below ranges:
* Neutrophil count < 1000/mm3
* Platelet count < 100,000/mm3L
* Hemoglobin < 9 g/dL (transfusion to meet eligibility allowed)
* AST/SGOT and ALT/SGPT > 3.0x upper limit of normal (ULN) without disease involvement or > 5.0x ULN if the transaminase elevation is due to disease involvement
* Alkaline phosphatase > 5.0x ULN without known bony metastases
* Serum bilirubin > 1.5x ULN
* Serum creatinine > 1.5x ULN or 24-hour creatinine clearance < 30 mL/min per Cockroft- Gault equation
* Total serum calcium < lower limit of normal (LLN) or if calcium is below LLN the corrected calcium for serum albumin is > LLN
* Serum potassium < 3.0
* Serum sodium < 130
* Serum albumin < 2.5 g/dL
* History of myocardial infarction. unstable angina, stroke or transient ischemic attack within 6 months prior to Day 1
* History or drug induced pneumonitis (both pembrolizumab and palbociclib can cause pneumonitis)
* Subjects requiring hemodialysis
* Patients with severe hepatic impairment (Childs-Pugh Class C).
* Other concurrent severe and/or uncontrolled medical conditions in the opinion of the investigator which will preclude participation
* Pregnancy (positive pregnancy test) or lactation
* Concomitant use of any other anti-cancer therapy or radiation therapy of the target lesion. Palliative radiation therapy is permitted to non-target lesions.
* Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) and adverse events (AEs) per CTCAE v5 | The dose limiting toxicity period is 4 weeks after starting the first dose of pembrolizumab
  Confirm the safety of the combination of Palbociclib and pembrolizumab in sarcomas for which PD-1 inhibitors are approved as defined by the incidence of DLTs

SECONDARY OUTCOMES:
Response rate per RECIST 1.1 criteria | 8 weeks following treatment intiation
  To assess the response (per RECIST 1.1 criteria) of patients with advanced UPS with the combination of CDK4/6 inhibitor and anti-PD-1 immunotherapy

OTHER OUTCOMES:
Progression free survival | Up to two years following completion of treatment
  To assess progression free survival as calculated by the time from start of treatment until the time of progression of disease or death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: John Rieth, MD, Principal Investigator — University of Iowa Hospitals & Clinics
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No